CLINICAL TRIAL: NCT04163939
Title: A Randomized Controlled Trial of Collar Use for Cervical Radicular Pain
Brief Title: Collar Use for Cervical Radicular Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: Synovation Medical Group (Other)
Responsible Party: Principal Investigator, Alexios Carayannopoulos, Medical Director, Comprehensive Spine Center; Chief of Physical Medicine and Rehabilitation Medicine, Chief of Lifespan Physican Group, Rhode Island Hospital, Newport Hospital, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1426278
Record Dates: First submitted 2019-11-01; First posted 2019-11-15 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Cervical Radiculopathy
Keywords: Neck pain
MeSH Terms: conditions — Radiculopathy; Neck Pain

STUDY DESIGN:
Intervention Model Description: To evaluate the effectiveness of treatment with Vista Therapy Collar for indication of cervical radicular pain, defined as pain radiating into one or both upper extremities compared to standard care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collar (Experimental): This group will wear a cervical collar for at least 30 minutes per day, 5 out of 7 days of the week
  Interventions: Other: Vista Therapy Collar
- Control (Placebo Comparator): This group will not wear the cervical collar
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Vista Therapy Collar — The patient will wear the cervical collar
  Arms: Collar
Other: Placebo — The patient will not wear the cervical collar
  Arms: Control

SUMMARY:
To evaluate the effectiveness of treatment in subjects with cervical radicular pain with Vista Therapy Collar, using a Visual Analog Scale, a Neck Disability Index and the SF-36 quality of life survey.

DETAILED DESCRIPTION:
To evaluate the effective of treatment with Vista Therapy Collar for indication of cervical radicular pain, defined as pain radiating into one or both upper extremities compared to a 'wait and see' approach.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years
2. Cervical radicular pain as defined by neck pain radiating to one arm with at least one of the following:

   * Provocation by neck movements or sensory changes in one or more adjacent dermatomes or diminished deep tendon reflexes in the affected arm.
   * Muscle weakness in one or more adjacent myotomes.
3. Neck Disability Index (NDI) score >= 10 points
4. VAS for neck pain >= 40
5. Subject has signed and dated the Patient Informed Consent /Patient Information Sheet prior to any study-related activities being conducted
6. Subject is willing and able to attend visits as scheduled and to comply with the study protocol

Exclusion Criteria:

1. Serious somatic or psychiatric disorder
2. Previous Neck Surgery
3. Whiplash as the primary incident
4. History of spinal tumor or infection
5. Cervical Instability per opinion of PI
6. Morbid Obesity (BMI>40)
7. TMJ issues
8. Subject is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound the results of this study
9. Subject is involved in current litigation regarding neck pain or injuries associated with neck pain
10. Subject is involved in Worker's Compensation litigation
11. Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | 90 days
  Questionnaire used to measure how neck pain affects activities of daily living. Each of the 10 items are scored from 0-5, the maximum score is 50. Higher scores signify greater disability. A score over 34 signifies complete disability.
SF-36 Quality of Life Survey | 90 days
  Questionnaire used to measure quality of life. All questions are scored on a scale from 0 to 100, with 100 representing the highest level of functioning possible. The total score is calculated as a percentage of the total points possible. A higher total percent signifies better outcomes.
Visual Analog Scale (VAS) | 90 days
  Scale used to measure pain. The subject will mark their pain on a scale with a length of 100mm. The scale is scored by measuring (mm) from the left end of the scale to the subject's marking. The VAS is scored from 0-100, higher scores signify a greater amount of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Comprehensive Spine Center, Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No